CLINICAL TRIAL: NCT03139968
Title: Reduction of the Operator's Radiation Exposure During CAG and PCI With RADPAD, a Randomized Controlled Double-blinded Trial
Brief Title: Reduction of Catheterization Radiation Exposure Pad
Acronym: RECAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: J.P.S Henriques (Other)
Responsible Party: Sponsor-Investigator, J.P.S Henriques, Prof. dr. J.P.S. Henriques, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECAP-RCT
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Radiation; Exposure Occupational; Coronary Interventions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient, operator and investigator are blinded to dummy drape vs RADPAD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiation absorbing drape (Experimental): Conventional protection measurements. Additionally, a lead-free protective, disposable drape containing bismuth and antimony (RADPAD®) is placed onto the sterile drape on the patient between the operator and the image intensifier.
  Interventions: Device: (sham) radiation absorbing drape (RADPAD®)
- Dummy group (Active Comparator): Conventional protection measurements. Additionally, a dummy, silicone, disposable drape (appearing identical to the experimental arm) is placed onto the sterile drape on the patient between the operator and the image intensifier.
  Interventions: Device: (sham) radiation absorbing drape (RADPAD®)
- Control goup (No Intervention): Only conventional protection measurements.

INTERVENTIONS:
Device: (sham) radiation absorbing drape (RADPAD®)
  Arms: Dummy group; Radiation absorbing drape

SUMMARY:
The RECAP-trial is a randomized controlled, double blinded, superiority trial studying the efficacy of the RADPAD®, a protective drape, that potentially reduces the scattered radiation received by the operator during diagnostic angiograms and percutaneous coronary interventions.

DETAILED DESCRIPTION:
A total of 750 consecutive diagnostic angiograms and percutaneous coronary interventions were randomly assigned to the radiation-attenuating (RADPAD®), a dummy drape or a control group in a 1:1:1 ratio. The drapes will be used in addition to conventional shielding material. Primary radiation exposure is measured blindly by a dose aware meter (Philips) positioned at a set location on the operator. Radiation exposure is measured by the X-ray systems (DAP in Gy·cm2). The primary outcome is the effective dose received by the first operator (mSv/Gy·cm2).

ELIGIBILITY:
Inclusion Criteria:

* All CAGs and PCI's

Exclusion Criteria:

* Other interventional procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Primary operator radiation exposure (mSv) | immediately post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vlastra W, Delewi R, Sjauw KD, Beijk MA, Claessen BE, Streekstra GJ, Bekker RJ, van Hattum JC, Wykrzykowska JJ, Vis MM, Koch KT, de Winter RJ, Piek JJ, Henriques JPS. Efficacy of the RADPAD Protection Drape in Reducing Operators' Radiation Exposure in the Catheterization Laboratory: A Sham-Controlled Randomized Trial. Circ Cardiovasc Interv. 2017 Nov;10(11):e006058. doi: 10.1161/CIRCINTERVENTIONS.117.006058. PMID 29089313